CLINICAL TRIAL: NCT04642339
Title: Randomized, Double-blind, Placebo Controlled, Clinical Trial of the Immunogenicity, Safety, and Efficacy of the Gam-COVID-Vac Combined Vector Vaccine in Prophylactic Treatment for SARS-СoV-2 Infection
Brief Title: Clinical Trial of the Immunogenicity, Safety, and Efficacy of the Gam-COVID-Vac Vaccine Against COVID-19 in Venezuela
Acronym: VENEZUELA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Ministerio del Poder Popular para la Salud de la República Bolivariana de Venezuela (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01V-Gam-COVID-Vac-2020
Record Dates: First submitted 2020-11-16; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: vaccine; COVID-19; adenoviral vector; SARS-CoV-2; Ad26; Ad5; Heterologous prime-boost vaccination
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5 | interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Gam-COVID-Vac (Experimental): Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2 infection
  Interventions: Biological: Gam-COVID-Vac
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Gam-COVID-Vac — Gam-COVID-Vac combined vector vaccine, 0,5ml/dose+0,5 ml/dose prime-boost immunization with component I (rAd26-S) and component II (rAd5-S) with 21 days interval
  Other Names: Sputnik V
  Arms: Vaccine Gam-COVID-Vac
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo controlled clinical trial of immunogenicity, safety and efficacy of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection in adults.

DETAILED DESCRIPTION:
Randomized, double-blind (blinded for trial subject and the study physician), placebo controlled clinical trial in parallel assignment of the immunogenicity, safety, and efficacy of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection in adults.

The trial will include 2,000 volunteers over the age of 18. After screening, they will be randomised (3:1) into two groups - a reference group of 500 volunteers who will receive the placebo and a study group of 1,500 volunteers who will receive the combined Gam-COVID-Vac vaccine against SARS-induced coronavirus infection-СoV-2oV-2. The trial subjects will be randomized into five age strata: 18-30, 31-40, 41-50, 51-60 and 60+ years. Each subject will participate in the trial for 180±14 days after the first dose of the study drug/placebo and will have one screening visit and five on-site visits to the study physician during the said period. The study drug/placebo will be administered intramuscularly during vaccination visits 1 and 2 (day 1 and day 21±2). Follow-up visits Nos. 3, 4, 5 will be conducted on days 28±2, 42±2 and 180±14, respectively. Blood samples will be taken from certain subjects during the following visits to assess the immunogenicity parameters on days 1, 42±2 and 180±14. During observation visits, vital indicators will be assessed on all trial subjects and changes in the subjects' condition and well-being will be recorded, observational visits may be remote, using telemedicine (TM) technologies. Additionally, the trial subjects will be able to have remote consultations with the study physician through the TM. Data from trial subjects will be collected through electronic case report forms.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of a subject to participate in the trial
2. Males and females aged 18+
3. Negative HIV, hepatitis, and syphilis test results
4. A negative test result for the presence of IgM and IgG antibodies to SARS CoV2 by enzyme immunoassay
5. A negative test result for COVID-2019 by PCR at screening visit
6. No COVID-2019 in the medical history
7. No contact with COVID-2019 persons within at least 14 days before the enrollment (according to trial subjects)
8. Consent to use effective contraception methods during the trial
9. Negative urine pregnancy test at the screening visit (for child-bearing age women)
10. Negative drugs or psychostimulants urine test at the screening visit
11. Negative alcohol test at the screening visit
12. No evident vaccine-induced reactions or complications after receiving immunobiological products in the medical history
13. No acute infectious and/or respiratory diseases within at least 14 days before the enrollment.

Exclusion Criteria:

1. Any vaccination/immunization within 30 days before the enrollment;
2. Steroids (except hormonal contraceptives) and/or immunoglobulins or other blood products therapy not finished 30 days before the enrollment.
3. Immunosuppressors therapy finished within 3 months before the enrollment
4. Pregnancy or breast-feeding
5. Acute coronary syndrome or stroke suffered less than one year before the enrollment
6. Tuberculosis, chronic systemic infections
7. Drug allergy (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, serum disease), hypersensitivity or allergic reaction to immunobiological products, known allergic reactions to study drug components, acute exacerbation of allergic diseases on the enrollment day
8. Neoplasms in the medical history.
9. Donated blood or plasma (450+ ml) within 2 months before the enrollment
10. Splenectomy in the medical history
11. Neutropenia (absolute neutrophil count <1,000 mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin <80 g/L), immunodeficiency in the medical history within 6 months before the enrollment
12. Active form of a disease caused by the human immunodeficiency virus, syphilis, hepatitis B or C
13. Anorexia, protein deficiency of any origin
14. Big-size tattoos at the injection site (deltoid muscle area), which does not allow assessing the local response to the study drug/placebo administration
15. Alcohol or drug addiction in the medical history
16. Participation in any other interventional clinical trial.
17. Any other condition that the study physician considers as a barrier to the trial completion as per the protocol
18. Study center staff and other employees directly involved in the trial and their families.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 42 day, 180 day
  Percentage of trial subjects with fourfold or more increase in the titer of SARS-CoV-2 glycoprotein-specific antibodies in 2,000 trial subjects on the drug administration day before injecting the first dose of the study drug/placebo and 42±2 and 180±14 days after the first dose

SECONDARY OUTCOMES:
Incidence and severity of adverse events | through the study (till day 180)
  Incidence and severity of adverse events in trial subjects within 6 months after injecting the first dose of the study drug/placebo
Virus-neutralizing antibody levels against the SARS-CoV-2 | 42 day
  Geometric mean virus-neutralizing antibodies titer in 500 trial subjects on the drug administration day before injecting the first dose of the study drug/placebo and 42±2 days after the first dose
Antibody levels against the SARS-CoV-2 glycoprotein | 42 day, 180 day
  Geometric mean titer of the SARS-CoV-2 glycoprotein-specific antibodies in 2,000 trial subjects on the drug administration day before injecting the first dose of the study drug/placebo and 42±2 and 180±14 days after the first dose
Percentage of trial subjects with coronavirus disease 2019 (COVID-19) | through the study (till day 180)
  Percentage of trial subjects with coronavirus disease 2019 (COVID-19) developed within 6 months, as confirmed with the method of polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis H García Piñero, MD, Principal Investigator — Children's Cardiology Hospital "Dr. Gilberto Rodriguez Ochoa"

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franco C, Cornejo A, Rodriguez M, Garcia A, Belisario I, Mayora S, Garzaro DJ, Jaspe RC, Hidalgo M, Parra N, Liprandi F, Zambrano JL, Rangel HR, Pujol FH. Sputnik V-Induced Antibodies against SARS-CoV-2 Variants during the Dissemination of the Gamma Variant in Venezuela. Viruses. 2024 Sep 18;16(9):1480. doi: 10.3390/v16091480. PMID 39339956